CLINICAL TRIAL: NCT03991663
Title: Prospective Cohort Study for Azoospermia Patients in Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD)
Brief Title: Azoospermia Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-azoospermia cohort
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Healthy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, semen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prospective Cohort Study for Azoospermia Patients was set up to investigate the short- and long-term health consequences in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, China.

DETAILED DESCRIPTION:
Infertility is an important problem with a multifactorial etiology that affects approximately 15% of couples who attempt pregnancy. Its cause in approximately 50% of infertile couples is male factors. Spermatogenesis is an extremely complex cell differentiation process involving 2,300 genes that regulate germ cell development and maturation.

Since last decade, Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD) has been used in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, and Henan Province Key Laboratory for Reproduction and Genetics. Information of patients (POI, PCOS, Endometriosis, azoospermia, ect) were recorded comprehensively. The current project plans to recruit azoospermia participants in our center. Biological samples, questionnaires and short/long term health data will be collected. The study is aimed to provide evidence for azoospermia prognosis.

ELIGIBILITY:
Inclusion Criteria:

* at least three semen evaluations performed on separate occasions, when the seminal specimen after centrifugation showed no sperm under the microscope and was then diagnosed according to several clinical parameters；

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: At least three semen evaluations performed on separate occasions, when the seminal specimen after centrifugation showed no sperm under the microscope and was then diagnosed according to several clinical parameters
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of serum FSH (Follicle stimulation hormone) | From date of inclusion, assessed by each 12 month, up to 40 years
  mIU/mL
Level of serum LH (luteinizing hormone) | From date of inclusion, assessed by each 12 month, up to 40 years
  mIU/mL
Level of serum T (Testosterone) | From date of inclusion, assessed by each 12 month, up to 40 years
  ng/ml

SECONDARY OUTCOMES:
Volume of testicles | From date of inclusion, assessed by each 12 month, up to 40 years
  Record the Length (mm)*Width (mm) of each testicle

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Background] Enatsu N, Chiba K, Fujisawa M. The development of surgical sperm extraction and new challenges to improve the outcome. Reprod Med Biol. 2015 Nov 27;15(3):137-144. doi: 10.1007/s12522-015-0228-2. eCollection 2016 Jul. PMID 29259430
- [Background] Deruyver Y, Vanderschueren D, Van der Aa F. Outcome of microdissection TESE compared with conventional TESE in non-obstructive azoospermia: a systematic review. Andrology. 2014 Jan;2(1):20-4. doi: 10.1111/j.2047-2927.2013.00148.x. Epub 2013 Nov 6. PMID 24193894